CLINICAL TRIAL: NCT01309503
Title: Speech Intelligibility in Noise and Estimation of Binaural Benefits Using the Hearing in Noise Test (HINT). Studies on Normal Hearing Children and Adults, Groups of Hearing Aid Users and Cochlea Implant Users.
Brief Title: Speech Intelligibility in Noise Using the Hearing in Noise Test (HINT)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Oslo University Hospital (Other)
Collaborators: University of Oslo (Other)
Responsible Party: Marte Myhrum, Master of Science in Electrionics, Signal processing., Oslo University Hospital
Other Study IDs: 2010/743a (REK )
Record Dates: First submitted 2011-03-03; First posted 2011-03-07 (Estimated); Last update posted 2011-03-29 (Estimated); Status verified 2011-03

CONDITIONS: Speech Intelligibility
MeSH Terms: conditions — Speech Intelligibility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Normal hearing: Children and adults
- Unilateral hearing loss
- Severe hearing loss high frequencies
- Adult CI users: Unilateral and bilateral CI
- Bilateral CI users: Children and adults
  Sequential CIs
  Simultaneous CIs

SUMMARY:
The main purpose of the study is to estimate speech intelligibility in noise. A Norwegian Hearing in Noise Test (HINT) for children will be implemented, and test results for normal hearing (NH) children and adults will be collected. Test results for groups of hearing aid (HA) users and test results for cochlea implant (CI) users will be collected and compared to the NH group and between groups of HA users and CI users. A group of single sided hearing loss patients will also be included. Binaural benefits of two ears, two HAs and two CIs will be estimated.

ELIGIBILITY:
Inclusion Criteria for the different groups:

1. Normal hearing group (note that some subjects are already recruited in the normal hearing group):

   * audiometric thresholds less than or equal to 25 dB HL for octave frequencies between 250 Hz and 8000 Hz
   * Adults between age 18 and 50 years
   * Children at different age groups between 6 and 12 years old
2. Unilateral hearing loss group

   * Single-sided hearing loss.
   * Using hearing aid or willing to try hearing aid on the side with hearing loss to estimate a potential binaural benefit with hearing aid.
   * Unilateral hearing loss inclusion criteria is thresholds within 25 dBHL and 70 dBHL for frequencies {125,250,500} Hz. Inclusion region increasing linearly with octave frequency to 40 dBHL and 95 dBHL for frequency 8000Hz. In addition a single threshold outside this hearing threshold inclusion region is accepted.
   * Contralateral normal hearing with audiometric thresholds less than or equal to 25 dB HL for octave frequencies between 250 Hz and 8000 Hz
3. Group with Severe hearing loss at high frequencies

   - Inclusion criteria is bilateral hearing loss within hearing levels where frequencies below 750 Hz can be normal or elevated down to 65 dBHL, for frequencies 1000 Hz and 1500 Hz all HL thresholds are accepted, frequencies 2000 Hz and above have threshold criteria 85 dBHL or above.
4. Adult CI users with unilateral and bilateral CI

   * All adult patients will be tested to the level of their performance.
   * HINT SRTs will be collected if HINT score in quiet is above 70%.
5. Bilateral CI users (Children)

   1. Sequential CIs group

      * Children that has got two CIs in two different operations, and operations are not within one year.
      * Inclusion of some of the patients participating in another ongoing sequential CI-study at the ENT department,and who has a HINT score above 70% in quiet. The requirement of a quiet percentage score above 70% is due to the bilateral benefit testing/estimation.
   2. Simultaneous CIs group

      * All children that has got two CIs in the same operation or sequentially within one year.
      * Children older than 6 years old.
      * Children as young as 5.5 years old can be included if they are considered ready for extended HINT testing.

Exclusion Criteria:

* None

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients at the ENT department, Oslo University hospital, Rikshospitalet. Normal hearing group recruited from different schools and kindergartens.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2011-03; Primary Completion 2014-03 (Estimated); Study Completion 2015-03 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Marte Myhrum, M.Sc., Principal Investigator — Oslo University Hospital; Greg Jablonski, PhD, Study Chair — Oslo University Hospital
Locations (1):
- Oslo university hospital, Oslo, Norway